CLINICAL TRIAL: NCT01578382
Title: Pathophysiology of Martorell Hypertensive Ischemic Leg Ulcer (HYTILU): A Comparison of Martorell HYTILU, Calciphylaxis and Venous Ulcer (Control)
Brief Title: Pathophysiology of Martorell Hypertensive Ischemic Leg Ulcer (HYTILU)
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: KEK-ZH-NR2010-0433/0
Record Dates: First submitted 2011-05-02; First posted 2012-04-16 (Estimated); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Hypertensive Ischemic Leg Ulcer; Calciphylaxis
Keywords: Martorell hypertensive ischemic leg ulcer; Calciphylaxis (calcific uremic arteriolopathy); Ischemic subcutaneous arteriolosclerosis; Hypertension; Diabetes; Medial calcinosis; Wound healing
MeSH Terms: conditions — Calciphylaxis; Hypertension; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood serum (2 tubes); blood plasma in citrate (2 tubes); blood plasma in heparin (2 tubes) Diseased skin tissue in formalin for paraffin embedded H-E histology; Diseased skin tissue snap frozen Diseased skin tissue in "RNA later" tube (1 tube)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Hypertensive ischemic leg ulcer: Twenty consecutive patients with Martorell HYTILU as defined in:
  Arch Dermatol 2010;146:961-968
- Calciphylaxis: Ten subjects with calciphylaxis (calcific uremic arteriolopathy) as described in:
  Vasa 1998;27:137-143
- Venous ulcer (controls): Twenty subjects with venous ulcers (CEAP C4-6) as described in:
  J Vasc Surg. 2004 Dec;40(6):1248-52

SUMMARY:
Martorell hypertensive ischemic leg ulcer is a severe type of skin necrosis (skin infarction) which occurs in long-term hypertensive subjects.

Calciphylaxis (calcific uremic arteriolopathy) is a severe type of skin necrosis (skin infarction) which occurs in subjects with end-stage kidney disease or after kidney transplantation.

DETAILED DESCRIPTION:
Comparative study including

* 20 consecutive patients with Martorell HYTILU
* 10 consecutive patients with Calciphylaxis (calcific uremic arteriolopathy)
* 20 patients with venous ulcer

The following parameters are measured in the blood serum:

White blood count; c-reactive protein; creatinine; calcium (total); free (ionized) calcium; phosphate; albumin; 25-hydroxyvitamin-D; 1-25-dihydroxyvitamin-D; homocysteine; cystatin C alphafetoin, osteoprotegerin; fibroblast growth factor 23 (FGF-23); globular arrest 1 (GLA-1)

The following parameters are measured in samples of diseased (necrobiotic) skin:

alphafetoin, osteoprotegerin; fibroblast growth factor 23 (FGF-23); globular arrest 1 (GLA-1)

ELIGIBILITY:
Inclusion Criteria:

* Having Martorell hypertensive ischemic leg ulcer (as defined above) or
* Having Calciphylaxis (calcific uremic arteriolopathy (as defined above) or
* Having a venous ulcer (as defined above)

Exclusion Criteria:

* None

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: n=20: Having Martorell hypertensive ischemic leg ulcer (as defined above) or n=10: Having Calciphylaxis (calcific uremic arteriolopathy (as defined above) or n=20: Having a venous ulcer (as defined above) (controls)
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2011-09; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Martorell HYTILU and calciphylaxis show both decreased tissue protection mechanisms against tissue calcification | 36 months
  Comparison of the calcification-protective factors GLA-1(serum protein alpha2-Heremans-Schmid glycoprotein/fetuin A), Osteoprotegerin, Fibroblast Growth Factor 23, and Alphafetoin in:
  * Martorell HYTILU (A1)
  * Calciphylaxis (calcific uremic arteriolopathy)(A2)
  * Venous ulcers (as control group)(B)

SECONDARY OUTCOMES:
Martorell hypertensive ischemic leg ulcer and calciphylaxis are both characterized by non-infectious inflammation | 36 months
  Comparison of C-reactive protein, procalcitonin and white blood cell count in:
  * Martorell HYTILU (A1)
  * Calciphylaxis (calcfic uremic arteriolopathy) (A2)
  * Venous ulcers (control group) (B)

CONTACTS AND LOCATIONS:
Overall Officials: Jürg Hafner, Professor, Principal Investigator — Department of Dermatology, University Hospital of Zurich, Switzerland
Locations (1):
- Department of Dermatology, University Hospital of Zurich, Zurich, Canton of Zurich, Switzerland